CLINICAL TRIAL: NCT06583616
Title: The Prognostic Value of Anion Gap in Predicting Mortality Among Patients With Acute Pulmonary Embolism
Acronym: PRAGUE-PE
Status: Recruiting | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Former of Head Cardiology Department, Universitas Diponegoro
Other Study IDs: Undip_Kardio_1
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Acute Pulmonary Embolism (PE)
Keywords: anion gap; acute pulmonary embolism; mortality
MeSH Terms: interventions — Acid-Base Equilibrium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survival Group: Patient with acute pulmonary embolism who survive after hospitalization
  Interventions: Diagnostic Test: Anion Gap

INTERVENTIONS:
Diagnostic Test: Anion Gap — Patient with acute pulmonary embolism who not survive after hospitalization

SUMMARY:
This study aims to evaluate the prognostic value of the anion gap in predicting mortality among patients with acute pulmonary embolism.

Researchers will collect information based on hospital registry as secondary data of in patient who had diagnosed as acute pulmonary embolism by using computed tomography scan (CT scan). The data consist of demographic data, clinical presentation, laboratory, and CT scan were collected from hospital registry by reviewing medical record. Then, the data was analyzed by using IBM SPSS Statistics v26.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 70 years old
* patient with acute pulmonary embolism

Exclusion Criteria -- patient with history of:

* heart failure
* valvular heart disease
* chronic obstructive pulmonary disease
* congenital heart disease
* sepsis
* chronic kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | During hospitalization, up to 1 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No